CLINICAL TRIAL: NCT06419114
Title: Exploration of Optical Coherence Tomography-Guided Transbronchial Biopsy in Peripheral Pulmonary Lesions
Acronym: OCTGTBIPPL
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Guanghong Zhou, Attending physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPHGZ01
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lung Neoplasm
Keywords: Peripheral Pulmonary Lesions
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biopsy specimen does not need to be extracted for DNA, and it is sent directly to the pathology department for examination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Coherence Tomography — Comparing the localization ability of OCT and R-EBUS in Peripheral Pulmonary Lesions and the predictive ability of lung cancer pathological classification
  Other Names: radial probe endobronchial ultrasound

SUMMARY:
In this prospective analysis, investigators collected and evaluated data from patients who underwent TBB at the Respiratory Endoscopy Center of Sichuan Provincial People's Hospital. The procedures utilized a novel approach combining OCT with R-EBUS for guidance. Eligibility for participation was determined based on established guidelines for the application of diagnostic flexible bronchoscopy in adults.

The admission criteria of this study were as followed: (1) voluntary participation and written informed consent signed, (2) age ≥ 18 years old, (3) the platelets count and PT, APTT tests were normal, (4) normal ECG, (5) found PPL's by chest computed tomography (CT) within 2 weeks and (6) could not detect the lesions through routine diagnostic bronchoscopy. The exclusion criteria of this study were as followed: (1) patients with contraindication of bronchoscopy (such as respiratory failure and acute cardio-cerebrovascular events), (2) patients who refuse biopsy because of physical reasons or personal wishes, (3) patients with the objective reasons (such as abundant blood supply around the lesion) who could not complete the biopsy, (4) patients who are participating in other clinical studies, (5) patients with poor compliance who are believed by the researchers to be unable to cooperate for the completion of the examination and follow-up, and (6) women who were pregnant.

R-EBUS and OCT In this study, all procedures were conducted using a standardized flexible bronchoscopy (Olympus, Japan) featuring an outer diameter of 4.2mm. R-EBUS system (Olympus, Japan) incorporated an ultra-thin radial ultrasonic probe (Olympus UM-S20-17S), which measures merely 1.4mm in diameter. The OCT (Yongshida Medical Technology, Guangdong, China) probe is a cylindrical catheter, 1.7mm in diameter and 150cm in length. Placing the probe through the working channel of bronchoscope for real time dynamic scanning of lesions.

Research Process In this study, the entirety of the procedures was performed by the same respiratory physician with 5 years of experience in respiratory endoscopic diagnosis and treatment, including preoperative evaluation, preparation, lesion localization and biopsy. The respiratory physician had examined the bilateral airways with flexible bronchoscopy after the completion of preoperative anesthesia and found no lesions. The subsequent step involved the precise placement of the OCT probe, guided by prior CT scan results. This stage was critical for marking the lesion, determining its nature (benign or malignant), and, in cases of malignancy, identifying its pathological classification. In instances where the OCT failed to identify any lesion, the R-EBUS was employed to facilitate lesion localization and biopsy. Conversely, when PPLs was detected via OCT, R-EBUS was additionally utilized to corroborate the PPLs localization and to assist in completing the biopsy procedure. For cases where OCT localization failed, R-EBUS would be used. After successful confirmation with R-EBUS, an attempt was made again to insert the OCT probe and completed biopsy. Rapid On-Site Evaluation (ROSE) was employed for the assessment of biopsy specimens. A total of five specimens were collected from each lesion and subjected to ROSE. In scenarios where ROSE provided a definitive diagnosis, no additional biopsies were deemed necessary. Conversely, in instances where ROSE yielded non-definitive results, further biopsy samples were obtained. All biopsy specimens were preserved in 10% formalin, preparing them for detailed histopathological analysis. The ultimate pathological diagnoses were determined based on the reports issued by the pathology department.

In this study, the demographics of all patients were documented, including age, gender, and smoking history. Additionally, detailed clinical parameters, such as the location and size of the lesions, airway grades (ranging from 0 to 24) that the PPLs located, location time of OCT and the number of specimens, were systematically recorded. investigators also conducted extensive follow-up to track histopathological outcomes, whether from surgical biopsies, CT-guided percutaneous transthoracic needle biopsies, or other diagnostic avenues, including chest CT performed two months post-procedure. All the patients were followed up by telephone or outpatient service on the 1st and 3rd day after the procedure, and adverse events were recorded. All individuals underwent general anesthesia and were fitted with a laryngeal mask.

DETAILED DESCRIPTION:
See details in"Brief summary"

ELIGIBILITY:
The inclusion criteria of this study were as followed: (1)Clinical diagnosis of PPL's by chest computed tomography (CT) within 2 weeks, (2)voluntary participation and written informed consent signed, (3) age ≥ 18 years old, (4) the platelets count and PT, APTT tests were normal, (5) normal ECG and (6) could not detect the lesions through routine diagnostic bronchoscopy. The exclusion criteria of this study were as followed: (1) patients with contraindication of bronchoscopy (such as respiratory failure and acute cardio-cerebrovascular events), (2) patients who refuse biopsy because of physical reasons or personal wishes, (3) patients with the objective reasons (such as abundant blood supply around the lesion) who could not complete the biopsy, (4) patients who are participating in other clinical studies, (5) patients with poor compliance who are believed by the researchers to be unable to cooperate for the completion of the examination and follow-up, and (6) women who were pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) voluntary participation and written informed consent signed, (2) age ≥ 18 years old, (3) the platelets count and PT, APTT tests were normal, (4) normal ECG, (5) found PPL's by chest computed tomography (CT) within 2 weeks and (6) could not detect the lesions through routine diagnostic bronchoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yield of OCT or R-EBUS-guided TBB in PPLs | baseline
  Ability to locate PPLs

SECONDARY OUTCOMES:
The pathological diagnostic value of OCT and R-EBUS | baseline
  The ability to distinguish between benign and malignant lesions and pathological classification of malignant lesions by using OCT and R-EBUS
The demographics of all patients | baseline and 2 months
  age(year), gender(male, female), and smoking history(yes or no)，the location and size of the lesions, airway grades (ranging from 0 to 24) that the PPLs located, location time(seconds) of OCT and the number of specimens(number=1,2,3...)，surgical biopsies, CT-guided percutaneous transthoracic needle biopsies, or other diagnostic avenues, including chest CT performed two months post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhou G, Yang Y, Liao Y, Chen L, Yang Y, Zou J. A pilot study of optical coherence tomography-guided transbronchial biopsy in peripheral pulmonary lesions. Expert Rev Med Devices. 2024 Sep;21(9):859-867. doi: 10.1080/17434440.2024.2389235. Epub 2024 Aug 6. PMID 39107968